CLINICAL TRIAL: NCT05990855
Title: Novel Methods to Increase Access and Facilitate Cognitive-behavioral Therapy for Insomnia in the Context of Depression: A Parallel-group Randomized Trial Comparing the Sleep Restriction Component Informed by Electroencephalography Measures to Sleep Restriction Based on Subjective Sleep Measures
Brief Title: Using Sleep Wearables to Adapt Cognitive-behavioral Therapy for Insomnia in the Context of Depression (CBTiA)
Acronym: CBTiA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Rébecca Robillard, Assistant Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022030
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Insomnia; Major Depressive Disorder; Persistent Depressive Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: All researchers involved in clinical assessments or data processing will be blinded to the assignment of these different conditions. Participants will be asked not to discuss the modality of sleep measurements (Sleep diary or EEG headband) with the research staff or their care provider.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCBTi-obj (Experimental): In the experimental condition, participants will complete a 5-week eCBTi program delivered via a mobile application while wearing an EEG headband (Muse S) during sleep. As part of the sleep restriction therapy component of CBTi, participants will be asked to follow an individualized sleep window (i.e., bed and wake schedule) which will be adjusted each week based on objective sleep data derived from their EEG recordings from the previous week. Participants will also receive a weekly sleep report based on this data.
  Interventions: Combination Product: eCBTi-obj
- eCBTi-subj (Active Comparator): In the active comparator condition, participants will complete the same 5-week eCBTi program, but will not be wearing an EEG headband during the intervention. As part of the sleep restriction therapy component of CBTi, participants will be asked to follow an individualized sleep window (i.e., bed and wake schedule) which will be adjusted each week based on the subjective sleep data derived from their sleep diary of the previous week, as is typically done during classical CBTi. Participants will not receive any EEG-based sleep report during the intervention.
  Interventions: Behavioral: eCBTi-subj

INTERVENTIONS:
Combination Product: eCBTi-obj — eCBTi based on objective sleep measures recorded by the Muse S headband.
  Arms: eCBTi-obj
Behavioral: eCBTi-subj — eCBTi based on standard subjective sleep measures recorded on the sleep diary.
  Arms: eCBTi-subj

SUMMARY:
This study aims to better adapt cognitive behavioral therapy for insomnia (CBTi) for people with comorbid depression by using objective sleep measures to tailor the behavioral interventions components of CBTi. Using ambulatory monitors, we also aim to investigate changes in brain activity and heart rate throughout the intervention. In this parallel-group randomized clinical trial, participants undergo one week of baseline ambulatory monitoring after which they are randomly assigned to one of two intervention arms: 1) digitally delivered CBTi (eCBTi) based on standard subjective sleep measures (sleep diary), or 2) eCBTi based on objective sleep measures (EEG headband). The intervention spans over 5-weeks, followed by a week of ambulatory monitoring and follow-up measures one week and one month after the end of the intervention. The study also includes a post-intervention interview to gather feedback on participant experiences. The overall protocol includes online questionnaires and structured clinical interviews assessing sleep, insomnia, and mental health, as well as treatment-related measures before, during, and after the intervention. It is anticipated that eCBTi using objective sleep measures will lead to better treatment acceptability, satisfaction, and effectiveness, including greater improvements in symptoms of insomnia and depression. It is also anticipated that sleep EEG and heart rate profiles will improve along the course of eCBTi.

DETAILED DESCRIPTION:
1. Background

   Insomnia is a major public health burden that disproportionately affects individuals with depression. Sleep disturbances are present in approximately 80-90% of cases of depression and are associated with more severe depressive symptoms, a less favorable prognosis, more medical and psychiatric comorbidities and a lower quality of life. Physiological hyperarousal, an abnormal state of increased responsiveness to stimuli marked by various physiological and psychological symptoms, is one of the pathophysiological mechanisms common to insomnia and depression. This state of hyperarousal is perceptible at the level of cortical activation and heart rate (HR) during sleep. Considering this overlapping of underlying mechanisms, intervening with sleep represents a promising way to simultaneously target cortical and cardiac hyperarousal, insomnia, and mood.

   CBTi is the recommended first line of treatment for chronic insomnia and is associated with significant improvement in depressive symptoms. CBTi is a multicomponent cognitive and behavioral treatment that targets the maladaptive thoughts and behaviors associated with the maintenance of insomnia. It includes five distinct intervention components, namely sleep hygiene education, cognitive therapy, relaxation training, stimulus control, and sleep restriction therapy.

   Sleep restriction therapy is one of the central components of CBTi which aims to restrict the time spent in bed according to a specific time window. This window is determined from the individual's sleep diary which is a subjective measure of sleep. As sleep estimation is particularly biased in those with insomnia and a depressive comorbidity, the use of sleep diaries is likely to increase stress and treatment-related burden as well as limit the accuracy of CBTi sleep manipulations. Another important limitation of CBTi in the context of psychiatric comorbidities is the high demand for this type of treatment in clinical settings coupled with the lack of trained clinicians which considerably restricts accessibility. The emergence of accurate ambulatory sleep monitors and of effective digitally delivered CBTi thus represents a new opportunity to increase access to CBTi, to anchor sleep restriction therapy on objective sleep measures and to observe changes happening at a physiological-level during treatment.

   To date, few studies have investigated the practical implications of wearable devices and digital technology in behavioral sleep medicine, especially with clinical populations. As highlighted in a recent systematic review, there is now a need to investigate whether the use of objective sleep data has the possibility to enhance the therapeutic outcomes associated with behavioral sleep interventions. A large clinical trial comparing treatment outcomes in users and non-users of wearable devices completing an eCBTi program showed similar treatment effects on insomnia symptoms. The authors concluded that the use of wearables may facilitate treatment for individuals who may have a difficult time completing daily sleep diaries. This has yet to be investigated in individuals with depression for whom sleep estimation represents an important struggle.
2. Objectives

   Primary aim:

   A) Evaluate if the use of objective sleep measures to adjust the sleep restriction window during CBTi enhances treatment acceptability, satisfaction, and effectiveness in people with insomnia and major depression;

   Secondary aims:

   B) Characterize the potential discrepancy between objective/subjective sleep measures in people with insomnia and major depression; C) Determine if the degree of discrepancy between objective/subjective sleep measures influences treatment acceptability, satisfaction, and efficacy; D) Characterize participant's experiences throughout the intervention and feedback about potential adaptations to better address challenges linked to insomnia treatment in the context of co-existing depression.

   E) Delineate how sleep EEG and HR profiles (measured prior to the intervention) relate to the nature and severity of depression and insomnia symptoms; F) Confirm the effects of eCBTi on the sleep EEG and HR indices linked to poor cardiovascular health, and mental health; G) Investigate the sleep EEG and HR correlates of eCBTi treatment response in terms of insomnia and depression symptoms; H) Identify potential physiological features in the EEG and HR profiles in pre-sleep wakefulness and during sleep that may be predictive of treatment response.
3. Methods

Participants will be allocated through randomization stratified by sex to one of two intervention arms: 1) eCBTi based on objective ambulatory sleep monitoring (eCBTi-obj) or 2) eCBTi based on subjective sleep diaries (eCBTi-subj; i.e. typical CBTi method). All intervention arms will be delivered as adjuncts to standard clinical care using the same smartphone application over a 5-week period. All researchers involved in psychiatric assessments will be blind to the intervention arms.

3.1 Recruitment, Consent, and Screening Recruitment will be achieved through institutional 'Permission to contact" registries, as well as through external recruitment with advertisements distributed via web-based platforms. Clinicians from affiliated institutions may also provide information about the study to their patients.

A research assistant will contact potential participants by email to send them a summary of the study and a link to complete an anonymous online screening form for the first set of eligibility criteria on a secured web platform (Qualtrics). The first question of this online form will ask participants to confirm they consent to take part to the screening process. This screening form will include the WHO-ASSIST item 2, Sleep Disorders Symptoms Checklist-25 (SDS-CL-25), Sleep Condition Indicator (SCI), Patient Health Questionnaire (PHQ-9). If the questionnaires indicate that the first set of eligibility criteria are met, the participant will be invited for the second and last screening step: a screening phone interview (based on the M.I.N.I.).

For participants found to be eligible after the screening phone interview, the research assistant will summarize the next steps of the study verbally and address any questions or concerns that participants may have at the end of the phone interview. Special care will be given to ensure that participants understand that their participation is entirely voluntary and that they can withdraw from the study at any stage. Eligible participants will be sent an electronic form containing the information and consent form (ICF). As part of that same electronic form, they will confirm consent by ticking consent boxes and entering their full name. Ongoing consent will also be obtained electronically at the follow-up time points.

3.2 Data collection and management

3.2.1. Baseline assessment Eligible participants will come on site to collect equipment to undergo 7-days of home-based ambulatory monitoring. They will return this equipment to the laboratory at the end of the week. The ambulatory equipment will include an EEG headband device (Muse S, InteraXon, Toronto, Canada) to be worn each night. They will also be lent a small sensor to be fixed on the abdomen using hypo-allergic tape to monitor skin temperature (i-button) and a Micro Motionlogger actigraphy watch, both to be worn across the 24-hour cycle for the entire duration of the week. During this period, participants will fill a daily sleep log (containing the core elements of the ''Consensus Sleep Diary''). Participants will be instructed on how to use this equipment on brief pre-recorded online videos.

On the seventh (last) day of the ambulatory monitoring period, participants will be asked to fill out a battery of questionnaires. This will inquire about general demographic and clinical information, sleep, daytime functioning, and mental health. They will also complete two 10-minute resting state EEG recordings from home: i) 30 minutes before sleep on the evening of the seventh day, and ii) 30 minutes after waking up on the following morning.

They will then return to the Sleep Research Unit to return the equipment and undergo further assessment with the Hamilton Depression Rating Scale (HDRS). They will be asked additional questions about the course of their mental disorders, including age at onset and duration of longest episode (inspired from the Diagnostic interview for genetic studies), as well as the proportion of time with depressive symptoms over the past 1, 5 and 10 years.

3.2.2. Experimental conditions Following baseline monitoring and questionnaires, participants will be randomly assigned to one of two intervention arms: eCBTi based on objective sleep measures (eCBTi-obj) or eCBTi based on standard subjective sleep measures (eCBTi-subj). The randomization process will be done by a computer-generated randomizer, stratified by sex. This will be managed by a research collaborator who will not be directly involved in clinical assessments or data processing. All researchers involved in clinical assessments or data processing will be blinded to the assignment of these different conditions.

The eCBTi intervention will be delivered from home across 5-weeks via the Insomnia Coach mobile application (U.S. Department of Veterans Affairs, Washington, USA). This eCBTi program is based on the CBTi Coach mobile application (U.S. Department of Veterans Affairs, Washington, USA) and the manual Cognitive Behavioral Therapy for Insomnia in Veterans. The mobile application contains all the standard CBTi interventions and includes reading material, auditory recordings, personalized feedback, as well as interactive components such as relaxation exercises and reminders.

Following the first intervention week, a sleep restriction window will be recommended for each participant. This sleep window will be determined based on the average total sleep time over the past week as recorded either by the Muse S Headband and scored by the automated scoring algorithm (eCBTi-obj group) or the sleep diaries (eCBTi-subj group). Following the initial sleep window recommendation, the sleep window will be adjusted weekly according to the past week's sleep efficiency (SE). If SE is equal to or above 90%, time in bed (TIB) will be increased by 15 minutes. If SE is between 85-89%, there will be no change to the prescribed sleep window for that week. If SE is below 85%, TIB will be decreased by 15 minutes. In all cases, the minimum sleep window will be 5 hours.

Throughout treatment, the eCBTi-obj group will wear the Muse S Headband and receive weekly feedback on their objective sleep data. Participants in the eCBTi-subj arm will not be wearing the headband and will be asked not to consult data from any other sleep monitor.

3.2.3. Follow-up measures Acceptability and satisfaction will be measured based on dropout rates. The day after the last intervention session, all participants will fill out, from home, a set of post-treatment questionnaires including questionnaires assessing treatment adherence (Modified Treatment Satisfaction Scale) and satisfaction (Treatment Component Adherence Scale) (about 1 hour). They will return to the Sleep Research Unit to undergo an in-person follow-up psychiatric assessment with the HDRS and a semi-structured exit interview to gather further insights (about 20 minutes). This will aim to gather feedback on participant's experiences throughout the intervention and potential adaptations to better address challenges linked to insomnia treatment in the context of co-existing depression. Before leaving the lab, participants will collect the equipment to complete another week of ambulatory monitoring from home with the Muse S Headband, iButton, Micro Motionlogger watch, and sleep log.

The questionnaires and HDRS will be repeated to evaluate sustained effects 1 week after the last day of intervention and 4 weeks after the last day of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years old
* Asymptomatic on the Sleep Disorders Symptoms Checklist-25 (except for insomnia)
* Symptomatic on the Sleep Condition Indicator (i.e. score above <3 on specific combination of items
* Current diagnosis of major depressive disorder or persistent depressive disorder confirmed by the Patient Health Questionnaire (PHQ-9) score > 10 and the MDE scale of the Mini International Neuropsychiatric Interview (M.I.N.I.)
* Having a smartphone and willingness to install a sleep intervention application on it

Exclusion Criteria:

* Current diagnosis of bipolar disorder, psychotic disorder or post-traumatic stress disorder confirmed by the M.I.N.I.
* Brain injury with loss of consciousness for over 5 minutes
* Self-reported substance use disorder (i.e. alcohol, cannabis, or illicit drugs) or > monthly use of illicit drugs reported on item-2 of the WHO Alcohol, Smoking and Substance Involvement Screening Test (except tobacco, alcohol, and cannabis)
* Body mass index > 45
* Shift work or rotating shifts within 1 month of study entry
* Recent travel to a difference time zone
* Any clinically significant cardiopulmonary, gastrointestinal, pancreatic, hepatic, renal, hematologic, endocrine, neurological (including seizure disorder), or sleep disorder (other than insomnia)
* Taking any psychotropic medications p.r.n. (If taking any antidepressant or sleep medications, needs to be on a stable dose for at least 1 month prior to study start).
* Taking stimulant medications including, but not limited to, Adderall, Concerta, Ritalin, Desoxyn, Dexedrine, Dextrostat, Ephedrine, Phentermine, Procentra, Vyvanse, and Selegline
* Insufficient English skills to provide informed consent, understand study instructions, or fill out questionnaires
* Individuals with mini-braids, dreadlocks, hair extension or natural afro-hair that can alter the EEG headband recording

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with treatment effectiveness as measured with the Modified Treatment Satisfaction Questionnaire for Medication | 7 weeks
  Satisfaction with treatment effectiveness, side effects, and convenience as rated on the Modified Treatment Satisfaction Questionnaire for Medication (mTQSM). The TQSM is a 14-item self-report scale with total scores ranging from 14-98, higher scores indicating greater treatment satisfaction. This questionnaire has been adapted for the purpose of this study: the term "medication" has been replaced by "intervention", and the term "condition" had been replaced by "symptoms of insomnia or depression".
Treatment acceptability as measured by the Treatment Acceptability/Adherence Scale | 7 weeks
  Adherence to CBT-I guidelines and perceived helpfulness of treatment guidelines as rated on the Treatment Acceptability/Adherence Scale (TAAS). The TAAS is a 10-item questionnaire with total scores ranging from 10-70, higher scores indicating greater treatment acceptability and adherence.

SECONDARY OUTCOMES:
Treatment acceptability as indexed by the number of drop outs | 7 weeks
  Acceptability as indexed by the number of drop outs in each intervention arm
Satisfaction with treatment effectiveness as measured by the Modified Treatment Satisfaction Scale | 7 weeks
  Perceived perceived symptom improvements as well as overall treatment satisfaction as measured by the Modified Treatment Satisfaction Scale (TSS). The TSS is a 7 item questionnaire with total scores ranging from 7 to 35, with higher scores indicating greater treatment satisfaction. In the present study, the TSS was adapted for insomnia to measure symptom improvement in key areas including insomnia, energy level, work productivity, coping, life enjoyment, hopefulness, self-esteem, and mood.
Changes in insomnia symptoms | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in insomnia symptoms as indicated by the Insomnia Severity Index-7 (ISI-7) total score from pre-intervention to the last follow-up time point after the end of the intervention. The ISI-7 is a 7 item questionnaire with total scores ranging from 0 to 28, with higher scores indicating more severe insomnia symptoms.
Changes in EEG-based sleep latency | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in EEG-based sleep onset latency from pre- to post-intervention.
Changes in EEG-based total sleep time | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in EEG-based total sleep time from pre- to post-intervention.
Changes in EEG-based slow wave sleep | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in the amount of slow wave sleep measured with the EEG headband from pre- to post-intervention.
Changes in EEG-based slow wave activity | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in the amount of slow wave activity (spectral power in the delta frequency range) from pre- to post-intervention.
Changes in EEG power spectra | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in global EEG power spectrum as measured by the EEG headband from pre- to post-intervention.
Changes in EEG-based slow wave morphometrics | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in the density, amplitude, rate of ascending/descending phases of sleep slow waves as measured by the EEG headband from pre- to post-intervention.
Changes in heart rate | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in heart rate measures including beats per minutes and heart rate variability from pre- to post-intervention.
Changes in subjective sleep quality | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in subjective sleep quality as rated by the subscales of the Leeds Sleep Evaluation Questionnaire (LSEQ): getting to sleep (GTS), quality of sleep (QOS), Awake following sleep (AFS), behaviour following wakening (BFW). The LSEQ is contains 10 items rated on a 10-cm line analogue scale. Scores for each item range from 0 to 10, with total scores ranging from 0-30 for the GTS and BFW subscales and from 0-20 for the QOS and AFS subscales. Higher scores indicate greater improvements in sleep. This will be measured from pre-intervention to the last follow-up time point after the end of the intervention.
Changes in subjective pre-sleep arousal | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in subjective pre-sleep arousal as rated on the Pre-Sleep Arousal Scale (PSAS) from pre- to post-intervention. The PSAS is a 16-item questionnaire with total scores ranging from 16 to 80, with higher scores indicating greater cognitive and somatic pre-sleep arousal.
Changes in unhelpful beliefs about sleep | From pre-intervention (week 0) to post-intervention (week 7)
  Changes in unhelpful beliefs about sleep as rated on the Dysfunctional Beliefs About Sleep (DBAS) questionnaire from pre- to post-intervention. The DBAS is a 16-item with total scores ranging from 0 to 160 and higher scores indicating greater dysfunctional beliefs and unrealistic expectations about sleep.
Changes in subjective fatigue | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in subjective fatigue as measured by the Fatigue Severity Scale (FSS) total score from pre-intervention to the last follow-up time point after the end of the intervention. The FSS is a 7 items scale with total scores ranging from 9 to 63, higher scores indicating greater fatigue severity.
Changes in clinician-assessed depression symptoms assessed with the Hamilton Depression Rating Scale | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in depression symptoms as assessed by the total score of the Hamilton Depression Rating Scale (HDRS). The HDRS is comprised of 17 items with total scores ranging from 0 to 52, with higher scores indicating greater depressive severity. This will be measured from pre-intervention to the last follow-up time point after the end of the intervention. Secondary analyses will be done on the HDRS total score minus the sleep items to disentangle the effects of sleep-related depression symptoms from that of other depression symptoms.
Changes in self-reported depression symptoms rated on the Quick Inventory of Depressive Symptomatology (QIDS). The QIDS is a 16-item questionnaire with total scores ranging from 0 to 27, with higher scores indicating greater depressive severity. | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in depression symptoms severity as assessed by the total score of the self-report version of the Quick Inventory of Depressive Symptomatology (QIDS). This will be measured from pre-intervention to the last follow-up time point after the end of the intervention. Secondary analyses will be done on the QIDS total score minus the sleep items to disentangle the effects of sleep-related depression symptoms from that of other depression symptoms.
Changes in self-reported depression symptoms rated on the Depression, Anxiety and Stress Scale | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in depression symptoms severity as assessed by the depression subscale of the Depression, Anxiety and Stress Scale (DASS-21) from pre-intervention to the last follow-up time point after the end of the intervention. The DASS-Depression subscale contains 7 items with total scores ranging from 0 to 42, and higher scores indicating greater symptom severity.
Changes in self-reported anxiety symptoms rated on the Depression, Anxiety and Stress Scale | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in anxiety symptoms severity as assessed by the anxiety subscale of the Depression, Anxiety and Stress Scale (DASS-21) from pre-intervention to the last follow-up time point after the end of the intervention. DASS-Anxiety subscale contains 7 items with total scores ranging from 0 to 42, and higher scores indicating greater symptom severity.
Changes in self-reported stress symptoms rated on the Depression, Anxiety and Stress Scale | From pre-intervention (week 0) to the last follow-up (week 10)
  Changes in stress symptoms severity as assessed by the stress subscale of the Depression, Anxiety and Stress Scale (DASS-21) from pre-intervention to the last follow-up time point after the end of the intervention. DASS-Stress subscale contains 7 items with total scores ranging from 0 to 42, and higher scores indicating greater symptom severity.
Objective-subjective discrepancy in sleep latency | 1 week
  Differences score where subjective sleep onset latency (derived from the sleep diary) is subtracted from objective sleep onset latency (derived by the EEG headband) collected at baseline (pre-intervention).
EEG-Actigraphy discrepancy in sleep latency | 1 week
  Differences score where actigraphy-based sleep onset latency is subtracted from EEG-based sleep onset latency collected at baseline (pre-intervention).
Objective-subjective discrepancy in total sleep time | 1 week
  Differences score where subjective total sleep time (derived from the sleep diary) is subtracted from objective total sleep time (derived by the EEG headband) collected at baseline (pre-intervention).
EEG-Actigraphy discrepancy in total sleep time | 1 week
  Differences score where actigraphy-based total sleep time is subtracted from EEG-based total sleep time collected at baseline (pre-intervention).
Objective-subjective discrepancy in sleep efficiency | 1 week
  Differences score where subjective sleep efficiency (derived from the sleep diary) is subtracted from objective sleep efficiency (derived by the EEG headband) collected at baseline (pre-intervention).
EEG-Actigraphy discrepancy in sleep efficiency | 1 week
  Differences score where actigraphy-based sleep efficiency (derived from the sleep diary) is subtracted from EEG-based sleep efficiency (derived by the EEG headband) collected in the entire sample at baseline (pre-intervention).
Qualitative feedback | 7 weeks
  Main themes emerging from qualitative interviews on participant's experiences with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rébecca Robillard, Principal Investigator — University of Ottawa Institute of Mental Health Research at The Royal
Locations (1):
- Sleep Research Unit, University of Ottawa Institute of Mental Health Research at the Royal, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Sharing of data outside of the primary institution leading the study such as through collaboration will be arranged only after express agreement with the PI.